CLINICAL TRIAL: NCT01369641
Title: A Pilot, Randomized, Self-controlled Study of the Effects of Intratympanic Sodium Thiosulfate on the Degree of Hearing Loss in Patients Receiving Cisplatin Therapy
Brief Title: The Effect of Sodium Thiosulfate Eardrops on Hearing Loss in Patients Who Receive Cisplatin Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 11D.99; 2011-03 (Other: CCRRC); JT 2092 (Other: JeffTrial Number)
Record Dates: First submitted 2011-06-07; First posted 2011-06-09 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: cisplatin; STS; sodium thiosulfate; Adults; dose range of 80-120mg/m2
MeSH Terms: conditions — Neoplasms | interventions — sodium thiosulfate; Sodium Chloride; Saline Solution; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Ear - Sodium Thiosulfate (STS) (Experimental): Subjects enrolled to study will have their ears randomized for treatment with STS. The experimental ear will receive STS treatments, while the comparator ear will receive a placebo.
  Interventions: Procedure: Insertion of Pressure Equalization (PE) Tubes; Drug: Sodium Thiosulfate (STS); Drug: Cisplatin
- Comparator Ear - Placebo (Placebo Comparator): Subjects enrolled to study will have their ears randomized for treatment with STS. The experimental ear will receive STS treatments, while the comparator ear will receive a placebo.
  Interventions: Procedure: Insertion of Pressure Equalization (PE) Tubes; Other: Saline (Placebo); Drug: Cisplatin

INTERVENTIONS:
Procedure: Insertion of Pressure Equalization (PE) Tubes — If the subject consents to participate in the study, a separate consent for insertion of pressure equalization (PE) tubes will be obtained. The PE tubes will then be inserted into the posterior inferior quadrant of the tympanic membrane in the office under topical anesthesia.
  Other Names: PE; tympanostomy tubes; myringotomy tubes
Drug: Sodium Thiosulfate (STS) — Drops of STS will be added to the experimental ear only prior to initial cisplatin infusion.
  Other Names: sodium thiosulphate
  Arms: Experimental Ear - Sodium Thiosulfate (STS)
Other: Saline (Placebo) — Drops of balanced saline solution will be added to the placebo comparator ear prior to initial cisplatin infusion.
  Other Names: saline solution
  Arms: Comparator Ear - Placebo
Drug: Cisplatin — Cisplatin chemotherapy infusion in the dose range of 80-120mg/m2
  Other Names: cisplatinum; cis-diamminedichloroplatinum(II); CDDP; Platinol; Platinol-AQ

SUMMARY:
This is a pilot, randomized, self-controlled study of the effects of intratympanic sodium thiosulfate (STS) on the degree of hearing loss in patients receiving cisplatin therapy. Sodium thiosulfate is an inactive ingredient contained in sulfacetamide ophthalmic solution which is used routinely as an otic solution delivered to the middle ear space.

The hypothesis of this study is that local administration of sodium thiosulfate (STS) will result in improved hearing compared to ears not receiving the study drug in patients receiving systemic cisplatin therapy.

DETAILED DESCRIPTION:
Platinum-based chemotherapeutic agents are used to treat a number of malignant tumors, both in children and adults. Examples of such tumors include: osteosarcoma, Wilms' tumor, rhabdomyosarcoma, neuroblastoma, Ewing's sarcoma, primary brain tumors, carcinoma, and various other solid tumors. Cisplatin is associated with a dose-dependent, high frequency sensorineural hearing loss. With increasing doses, the hearing loss worsens to include the speech frequencies. Vestibular function can also be damaged by platinum-based toxicity. Cisplatin causes ototoxicity through the formation of reactive oxygen species and activation of the apoptotic pathway in outer hair cells and the stria vascularis.

Rates of ototoxicity are approximately 80% with audiologic findings of hearing loss, and 20% with symptomatic hearing loss. These numbers are higher for those receiving high dose cisplatin, children, those with prior irradiation and those with prior hearing loss.

A number of agents have been investigated in animal models as otoprotection against the toxic effects of cis- and carboplatin. Among these, sodium thiosulfate (STS) has shown particular promise as an otoprotective agent. STS is approved by the US Food and Drug Administration (FDA) as an antidote for cyanide and nitroprusside toxicity and for calciphylaxis. STS has been shown to act as both an antioxidant as well as a chelating agent in vivo. The chelating properties of the sulfur-thiol functional group are believed to be responsible for the otoprotective effects of STS, binding to, and inactivating the platinum. The thiol compound may also act to scavenge reactive oxygen species produced by the platinum, thus preventing the initiation of the apoptotic pathway.

Several studies have demonstrated the otoprotective effects of intravenous STS in animal models. Subsequent studies have shown similar benefit when STS is administered intravenously to humans. A major drawback to this mode of delivery, however, is the fear that it reduces the anti-tumor activity of the platinum. Sodium thiosulfate is believed to bind to cisplatin, forming a complex that is then excreted by the kidneys. Though this may decrease the ototoxicity associated with the platinum, it may also decrease the anti-neoplastic properties of the agent. There are conflicting reports of reduced tumoricidal properties of STS in vitro, though there are no in vivo studies suggesting this adverse effect in vivo.

In view of the potential for systemic STS to reduce the tumoricidal effects of platinum agents, researchers have sought an alternate mode of delivery. Recent animal studies have examined the effect of sodium thiosulfate delivered locally to the middle ear space. Stocks, et al demonstrated an otoprotective effect of STS delivered to the middle ear space of guinea pigs. Wang, et al showed complete prevention of the ototoxic effects of cisplatin in guinea pigs treated with round window application of STS. In their study, both the compound action potential (CAP) and distortion product otoacoustic emissions (DPOAE) were unchanged, and both outer hair cells (OHC) and inner hair cells (IHC) were preserved. This effect, however, was not demonstrated in a similar study by Wimmer, et al. The temporal and spatial separation of the platinum and STS in these animal studies prompted Zuur and colleagues to state that, "in the future, it may be desirable to examine additional possibilities for two-route administration schemes for chemotherapy and otoprotective drugs in humans." There are no studies to date of intratympanic sodium thiosulfate in humans.

ELIGIBILITY:
Inclusion Criteria:

1. Adults receiving cisplatin therapy in the dose range of 80-120mg/m2
2. Subjects are capable of giving informed consent, or if appropriate, have an acceptable surrogate capable of giving consent on the subject's behalf.

Exclusion Criteria:

1. Subjects with active middle ear disease (unilateral or bilateral)
2. Subjects with prior treatment with platinum-based chemotherapeutic agent or other ototoxic agent
3. Subjects with an allergy to sodium thiosulfate
4. Subjects with tumors involving cranial nerve VIII
5. Subjects with preexisting absence of otoacoustic emissions (unilateral or bilateral)
6. Subjects with more than 5 dB interaural difference in puretone threshold on initial audiometric screening
7. Chronic use of known ototoxic agent (e.g. furosemide, aminoglycosides, etc)
8. Subjects with a history of prior irradiation to the head and neck.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-08-24 (Actual); Primary Completion 2013-03-10 (Actual); Study Completion 2013-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Cognetti, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospital — http://www.JeffersonHospital.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Sodium Thiosulfate (STS) Ear & Placebo Ear: Subjects enrolled to study will have their ears randomized for treatment with STS. The experimental ear will receive STS treatments, while the comparator ear will receive a placebo.
  Insertion of Pressure Equalization (PE) Tubes: If the subject consents to participate in the study, a separate consent for insertion of pressure equalization (PE) tubes will be obtained. The PE tubes will then be inserted into the posterior inferior quadrant of the tympanic membrane in the office under topical anesthesia.
  Sodium Thiosulfate (STS): Drops of STS will be added to the experimental ear only prior to initial cisplatin infusion.
  Cisplatin: Cisplatin chemotherapy infusion in the dose range of 80-120mg/m2
Period: Overall Study
Arm/Group | Sodium Thiosulfate (STS) Ear & Placebo Ear
Started | 1
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sodium Thiosulfate (STS) Ear & Placebo Ear
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.26 (0)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Intratympanic Sodium Thiosulfate (STS)
Description: To assess the efficacy of intratympanic sodium thiosulfate (STS) on reducing the degree or incidence of hearing loss in patients receiving systemic cisplatin therapy using puretone and speech audiometry, and distortion product otoacoustic emissions (DPOAE).
  Pure tone and speech audiometry: hearing will be assessed prior to any initiation of cisplatin therapy, again at three weeks, 6 weeks, 12 weeks, and every 6 months thereafter for up to one year.
Time Frame: Through 1 year post-treatment
Arm/Group | Sodium Thiosulfate (STS) Ear & Placebo Ear
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Sodium Thiosulfate (STS) Ear & Placebo Ear
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Thiosulfate (STS) Ear & Placebo Ear (N=1)
Ear infaction and tympanic perforation (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study terminated due to poor accrual, prior to subjects being analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes